CLINICAL TRIAL: NCT02226081
Title: Assessment of ShearWave™ Elastography in the Ultrasonic Diagnosis of Breast Cancer in Chinese Patients
Brief Title: ShearWave™ Elastography of Breast Lesions in Chinese Patients
Acronym: BE3
Status: Completed | Type: Observational
Sponsor: SuperSonic Imagine (Industry)
Responsible Party: Sponsor
Other Study IDs: BE3; ChiCTR-DDT-14004785 (Registry Identifier: China Clinical Trial)
Record Dates: First submitted 2014-08-25; First posted 2014-08-26 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Breast Neoplasms
Keywords: breast lesion; ultrasound; BI-RADS; women; malignancy
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
We aim to determine if adding ShearWave Elastography to a standard ultrasound breast exam can improve the characterization (classification) of breast lesions.

DETAILED DESCRIPTION:
Chinese women are known to have denser breasts than women in Western countries. Mammography cannot find abnormalities easily in denser breasts, while breast ultrasound is not affected by density. Adding elastography, a stiffness measurement, to a breast ultrasound exam should improve the diagnosis of a lesion.

ELIGIBILITY:
Inclusion Criteria:

* female
* 18 years of age or older
* known breast lesion that has not been managed or treated
* referred for a breast ultrasound because of a breast mass found on at least one of the following examinations:

  * physical palpation
  * mammography
  * ultrasound exam
  * MRI

Exclusion Criteria:

* Women who are unwilling or unable to provide informed consent
* Women with breast implants
* Women who are pregnant or breastfeeding
* Women in whom all lesions are diagnostically categorized as BI-RADS 0, 1 or 6
* Women with previous ipsilateral breast surgery
* Women with no visible breast mass on ultrasound examination
* Women with axillary metastatic lymph nodes only
* Women with foreign body in the breast
* Women who are not Chinese nationality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese women (age of majority) who have been referred to a hospital or clinical for a breast ultrasound evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 2273 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Increase in specificity of breast ultrasound imaging when considering stiffness measurements | Within 18 months of the study start date

SECONDARY OUTCOMES:
Change of sensitivity and negative predictive value of breast ultrasound imaging when considering stiffness measurements | Within 18 months of the study start date
Increase in positive predictive value for biopsy of breast ultrasound when considering stiffness measurements | within 18 months of the study start date

CONTACTS AND LOCATIONS:
Overall Officials: Cai Chang, Principal Investigator — Fudan University; Anhua Li, Principal Investigator — Sun Yat-sen University
Locations (22):
- China (22):
  - 1st Affiliated Hospital of PLAGH (304), Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - People's Liberation Army General Hospital (301), Beijing
  - Affiliated Hospital of Binzhou Medical University, Binzhou
  - Sichuan Provincial People's Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - Fujian Provincial Cancer Hospital, Fuzhou
  - Guangdong Provincial Traditional Chinese Medical Hospital, Guangzhou
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou
  - Sun-Yat Sen University Cancer Center, Guangzhou
  - 1st Affiliated Hospital of Harbin University, Harbin
  - Hefei 2nd People's Hospital, Hefei
  - Jiangsu Provincial Hospital, Nanjing
  - Yinzhou People's Hospital, Ningbo
  - Fudan University Cancer Center, Shanghai
  - 1st Affiliated Hospital of China Medical University, Shenyang
  - 4th Affiliated Hospital of China Medical University, Shenyang
  - Shengjing Hospital of China Medical University, Shenyang
  - General Hospital of TISCO, Taiyuan
  - Shanxi Dayi Hospital, Taiyuan
  - 1st Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - 1st Affiliated Hospital of Zhengzhou University, Zhengzhou

REFERENCES:
- [Result] Lin X, Chang C, Wu C, Chen Q, Peng Y, Luo B, Tang L, Li J, Zheng J, Zhou R, Cui G, Li A, Wang X, Qian L, Zhang J, Wen C, Gay J, Zhang H, Li A, Chen Y. Confirmed value of shear wave elastography for ultrasound characterization of breast masses using a conservative approach in Chinese women: a large-size prospective multicenter trial. Cancer Manag Res. 2018 Oct 11;10:4447-4458. doi: 10.2147/CMAR.S174690. eCollection 2018. PMID 30349377
- See also: Full-length article in Cancer Management and Research journal — https://www.dovepress.com/confirmed-value-of-shear-wave-elastography-for-ultrasound-characteriza-peer-reviewed-article-CMAR